CLINICAL TRIAL: NCT02238951
Title: Use of mHealth to Support Nurse-directed Care Coordination for Chemotherapy Patients: Improving Health, Healthcare Delivery, and Healthcare Utilization.
Brief Title: Cancer Care Coordination for Chemotherapy Patients
Acronym: 4CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: McKesson Foundation (Other); Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 551190
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Cancer
Keywords: care coordination, mobile health, chemotherapy, technology
MeSH Terms: conditions — Neoplasms | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile Health (mHealth) (Experimental): Care coordination using mHealth technology enhancements
  Interventions: Other: Mobile Health (mHealth)
- No mHealth (Active Comparator): Care coordination without mHealth enhancements
  Interventions: Other: No mHealth

INTERVENTIONS:
Other: Mobile Health (mHealth) — Participants receive care coordination throughout their chemotherapy treatment using mHealth technology
  Other Names: Android-based device; Mobile health; Patient Health Network
  Arms: Mobile Health (mHealth)
Other: No mHealth — Participants receive the same evidence-based care coordination without mHealth technology
  Arms: No mHealth

SUMMARY:
The purpose of this study is to compare nurse-led care coordination for persons receiving cancer chemotherapy treatment incorporating mobile health technology to nurse-led care coordination without any mobile health enhancements.

DETAILED DESCRIPTION:
This study will randomize sixty (60) participants receiving cancer chemotherapy treatment to receive nurse-led care coordination using a HIPAA-compliant mobile health platform compared to no technology-enhanced care coordination.

All participants receive nurse-led care coordination throughout chemotherapy treatment.

RESEARCH AIMS:

* Demonstration of a HIPAA-compliant social networking platform;
* Facilitate communication and collaboration among patients with cancer and their care team;
* Assess patient health outcomes (chemotherapy-related physical and psychological side effects; pain, quality of life and patient satisfaction)
* Assessment of healthcare utilization including emergency department visits, unplanned clinic visits and hospitalization;
* For patients assigned to the mobile health care coordination, understanding their experience of use of the technology

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Newly diagnosed cancer - any site or stage
* Initiating chemotherapy
* Ability to read and write English
* Manual dexterity sufficient to use a tablet technology
* Cognitive capacity to participate
* Preferential recruitment of publicly insured and/or living in rural communities

Exclusion Criteria:

* Oral chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Outcome | Baseline, 3 months, 6 months
  Pain

SECONDARY OUTCOMES:
Demonstration of a HIPAA-compliant platform to coordinate care overtime | Baseline, 6 months
  * Technology Usability and Acceptance
  * Patient engagement with technology
  * Use of electronic medical record features to communicate with providers

OTHER OUTCOMES:
Change in Patient Health Outcomes | Baseline, 3 months, 6 months
  * Treatment related symptoms
  * Psychological Distress
  * Quality of Life
Change in Healthcare Outcomes | Baseline, 6 months
  * Processes of care coordination
  * Patient engagement
  * Patient satisfaction
Change in Healthcare Utilization | Baseline, 3 months, 6 months
  * Emergency department visits
  * Unplanned hospitalizations
  * Unplanned clinic visits
Mobile health usability overtime | 2 weeks, 8 weeks
  Guided interviews with technology group to assess understanding and usability of the mobile technology platform to communicate and coordinate care

CONTACTS AND LOCATIONS:
Overall Officials: Jill G Joseph, MD, PhD, Principal Investigator — University of California, Davis Betty Irene Moore School of Nursing
Locations (1):
- UC Davis Comprehensive Cancer Care Center, Sacramento, California, United States